CLINICAL TRIAL: NCT04539717
Title: Abbreviated MRI for HCC Screening in Cirrhotic Patients (FAST-MRI Study)
Brief Title: FAST (Focused Abbreviated Screening Technique)-MRI Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, San Diego (Other); Duke University (Other); University of Wisconsin, Madison (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bachir Taouli, Professor, Radiology and Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 19-1409; 1R01CA249765-01 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC); Liver Cirrhosis
Keywords: Magnetic Resonance Imaging (MRI); Ultrasound (US); Liver Diseases; Elastography
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected to measure AFP, AFP-L3 and DCP (Des-carboxy-prothrombin), ctDNA and other tumor markers. The research team will not perform whole genome sequencing (i.e., sequencing of a human germline or somatic specimen with the intent to generate the genome or exome sequence of that specimen) as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to compare the diagnostic value of a reconstructed abbreviated Magnetic Resonance Imaging (MRI) from a full clinical exam, compared to ultrasound (US) for screening of liver cancer. Blood markers will be evaluated to determine their correlation to imaging. This study will help to determine whether abbreviated MRI is superior to ultrasound for diagnosis of liver cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fastest growing cause of cancer death in the United States and now kills over 30,000 Americans annually. To reduce the morbidity and mortality caused by this aggressive cancer, current practice guidelines recommend semi-annual abdominal ultrasound in adults with cirrhosis, the leading risk factor for HCC, to detect HCC nodules when they are small and treatable. Unfortunately, US has poor sensitivity for early-stage HCC in cirrhosis, failing to detect treatable cancer in over half of affected patients. Alternatives such as computed tomography (CT) or magnetic resonance imaging (MRI) are also not ideal due to ionizing radiation (CT), higher cost (MRI), or long exam time (~30-45 min for MRI). An optimal and fast HCC screening method is urgently needed and should be more sensitive and cost-effective than US and avoid ionizing radiation.

This is a prospective cross-sectional single arm non randomized multicenter study enrolling in 4 American centers as follows: Icahn School of Medicine at Mount Sinai-ISMMS, University of California San Diego-UCSD, University of Wisconsin-UW, and Duke University. The composite reference standard will incorporate the clinical results of the full baseline MRI exam and of subsequent imaging and pathology data collected over the next 6 months. Routine clinical follow-up imaging at 6 months will be observed. Patients will then be classified as positive for HCC, negative for HCC, or excluded.

ELIGIBILITY:
Inclusion Criteria

* Liver cirrhosis of any etiology.
* 18 years of age and older.
* Enrolled in screening/surveillance program for HCC.
* Clinically indicated imaging-based screening for HCC.
* Willing and able to complete all study procedures within specified time windows.
* Patient is able to give informed consent for this study.

Exclusion Criteria

* Contra-indications to MRI.
* Age less than 18 years.
* Patients with chronic renal failure or inability to tolerate contrast.
* Inability to undergo MRI due to lack of insurance coverage.
* Prior negative screening exam less than 5 months prior to enrollment.
* Prior hepatic resection.
* Post liver transplantation.
* Previously treated HCC or other liver neoplasm.
* Any other condition or factor that in judgment of study investigator may interfere with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed liver cirrhosis enrolled in imaging-based screening for HCC.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence of HCC | Within 6 months after initial index imaging (MRI & US)
  The presence of HCC will be determined by a composite reference standard. This composite reference standard incorporates the results of the complete MRI exam, pathology, and clinical follow-up.

SECONDARY OUTCOMES:
Circulating tumor DNA (ctDNA) | Within 1 year of blood processing
Serum AFP | Within 1 year of blood processing
  Serum Alpha-Fetoprotein
Cost-effectiveness | Within 1 year after initial index imaging (MRI & US).
  The cost-effectiveness will be assessed using a micro simulation model.

CONTACTS AND LOCATIONS:
Overall Officials: Bachir Taouli, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis S, Wildman-Tobriner B, Cuevas J, Calle S, Bolger I, Wang K, Joshi H, Mankowski Gettle L, Yang JD, Min JH, Sirlin CB, Reeder SB, Bashir MR, Taouli B. Quality of Gadoxetate-enhanced MRI versus US during Hepatocellular Carcinoma Screening in Participants with Cirrhosis. Radiology. 2026 Feb;318(2):e251497. doi: 10.1148/radiol.251497. PMID 41665498